CLINICAL TRIAL: NCT01970709
Title: DART Registry: Diagnosing Adverse Drug Reactions Registry
Brief Title: Diagnosing Adverse Drug Reactions Registry
Acronym: DART
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Renaissance RX (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Other Study IDs: 2013-101
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Genetics of Drug Metabolism
Keywords: Adverse Drug Reactions; Emergency Department Visits; Hospitalizations; Pharmacogenomic
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — Buccal swab
Oversight: Data Monitoring Committee: No

SUMMARY:
This multicenter Registry is to assess whether the use of pharmacogenomic data results in a meaningful change in a subject's drug or dose regimen. In addition, the Registry will evaluate the relationship between adverse drug reactions (ADR) and genotype and assess resource utilization (emergency department visits and hospitalizations) associated with ADR.

ELIGIBILITY:
Inclusion Criteria:

* Subject has care coordinated at the treating physician's outpatient clinic;
* Subject has provided written informed consent;
* Subject is taking at least three (3) regularly scheduled medications, excluding as needed (PRN) medications, over the counter medications and nutritional supplements; two (2) of which are known to be affected by genetic allelic variation.
* Subject's treating physician has a clinical suspicion that the subject is experiencing adverse signs or symptoms related to a prescribed medication or is not achieving the intended effect from the medication.

Exclusion Criteria:

* Subject has a history of chronic renal dysfunction, Chronic Kidney Disease Stage 4 or 5;
* Subject has a history of abnormal hepatic function within the last 2 years (INR >1.2 not attributable to anticoagulant medications, AST (aspartate aminotransferase) or ALT (alanine aminotransferase) >1.5x normal, or suspected cirrhosis);
* Subject has a history of malabsorption (short gut syndrome);
* Subject has a history of any gastric or small bowel surgery;
* Subject is currently hospitalized;
* Subject is currently being treated with intravenous medication;
* Subject underwent prior pharmacogenomic testing with results reported within the last 12 months.

Subjects may be eligible within 60 days from the date of pharmacogenomic testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects over the age of 18, taking three or more medications, two of which are metabolized by the CYP450 pathway.
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of meaningful change in drug regimen | 60 days
  The primary endpoint of the study is the binary occurrence of meaningful change in drug regimen, defined in each subject when:
  * A genotype known to affect a drug the subject is taking is identified, and
  * The subject's treating physician makes at least one drug regimen change in concordance with the PharmD recommendations.

SECONDARY OUTCOMES:
Change in the regimen of drugs controlled by genes of interest over the 12 months prior to enrollment and change in the regimen of drugs controlled by genes of interest over the 60 days following receipt of pharmacogenetic test results. | 60 days
Number of ADR per month over the 12 months prior to enrollment and number of ADR per month over the 60 days following receipt of pharmacogenomic test results. | 60 days
Frequency of genome-based PharmD recommendations to alter drug or dose. | 60 days
Emergency department visits and hospitalizations | 60 days
  Emergency department visits over the 12 months prior to enrollment, emergency department visits over the 60 days following receipt of test results, hospitalizations over the 12 months prior to enrollment, and hospitalizations over the 60 days following receipt of test results.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Edwards Lake Medical Center, Birmingham, Alabama
  - Gerald Harris MD, Glendale, Arizona
  - Holland Center for Family Health, Peoria, Arizona
  - AZ Pain Center, Phoenix, Arizona
  - Olga Voroshilovsky, Los Angeles, California
  - Institute for Regenerative Medicine and Clinical Research, Pasadena, California
  - Boulder Medical Center, Boulder, Colorado
  - Prime Healthcare - Anthony Roselli MD, Avon, Connecticut
  - Washington Pain Center, Washington D.C., District of Columbia
  - Continental Research Network, Doral, Florida
  - Latin Foundation for Health, Miami, Florida
  - Primary Care Associates, P.A., Stuart, Florida
  - Roman Medical Group, Columbus, Georgia
  - Wellness Medicine, Hampton, Georgia
  - Ocmulgee Physicians, Macon, Georgia
  - Macon Family Health Center Inc., Macon, Georgia
  - Your Personal Physician, Rome, Georgia
  - Valley Health Care, Rome, Georgia
  - Dr. B. Abraham PC, Snellville, Georgia
  - Candler Internal Medicine, Statesboro, Georgia
  - Primary Health Associates, Orland Park, Illinois
  - Women's Care Center, Lexington, Kentucky
  - Healthy Heart Cardiology, Grandville, Michigan
  - Heart Cardiology Consultants, Southfield, Michigan
  - Union Square Medical Associates, PC, Elizabeth, New Jersey
  - United Medical PC, Lyndhurst, New Jersey
  - Internal Medicine Specialists of Alamogordo, P.C., Alamogordo, New Mexico
  - Lovelace Rehabilitation Hospital, Albuquerque, New Mexico
  - Sage Neuroscience Center, Albuquerque, New Mexico
  - Geriatrics Associates, PAC, Albuquerque, New Mexico
  - Isabel C Vigil MD, Las Cruces, New Mexico
  - Larry F Berman MD PC, Charlotte, North Carolina
  - Lakewood Pediatrics and Family Medicine, Durham, North Carolina
  - Carolina Urology Partners, Gastonia, North Carolina
  - Carolina Neurosurgery and Spine Associates, Greensboro, North Carolina
  - Comprehensive Pain Center, Columbus, Ohio
  - Knightsbridge Internal Medicine and Cardiology Associates, Inc, Columbus, Ohio
  - Gateway Health and Wellness LLC, Columbus, Ohio
  - Robert E Barkett Jr MD, Mansfield, Ohio
  - Midwestern Internal Medicine Associates (MIMA), Marion, Ohio
  - Stonegate Family Health, Reynoldsburg, Ohio
  - Primary Care Associates - Unity, Tallmadge, Ohio
  - Easton Cardiovascular Associates, Easton, Pennsylvania
  - Carolina Center For Advanced Management Of Pain, Greenville, South Carolina
  - Colonial Family Practice, Sumter, South Carolina
  - Palmetto Adult Medicine, Sumter, South Carolina
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Mark A. Sanders, DO, Fort Worth, Texas
  - Emporia Medical Associates, Emporia, Virginia

REFERENCES:
- [Background] Onder G, Petrovic M, Tangiisuran B, Meinardi MC, Markito-Notenboom WP, Somers A, Rajkumar C, Bernabei R, van der Cammen TJ. Development and validation of a score to assess risk of adverse drug reactions among in-hospital patients 65 years or older: the GerontoNet ADR risk score. Arch Intern Med. 2010 Jul 12;170(13):1142-8. doi: 10.1001/archinternmed.2010.153. PMID 20625022
- [Background] Lazarou J, Pomeranz BH, Corey PN. Incidence of adverse drug reactions in hospitalized patients: a meta-analysis of prospective studies. JAMA. 1998 Apr 15;279(15):1200-5. doi: 10.1001/jama.279.15.1200. PMID 9555760
- [Background] Budnitz DS, Lovegrove MC, Shehab N, Richards CL. Emergency hospitalizations for adverse drug events in older Americans. N Engl J Med. 2011 Nov 24;365(21):2002-12. doi: 10.1056/NEJMsa1103053. PMID 22111719
- [Background] Mallet L, Spinewine A, Huang A. The challenge of managing drug interactions in elderly people. Lancet. 2007 Jul 14;370(9582):185-191. doi: 10.1016/S0140-6736(07)61092-7. PMID 17630042
- [Background] Epstein RS, Moyer TP, Aubert RE, O Kane DJ, Xia F, Verbrugge RR, Gage BF, Teagarden JR. Warfarin genotyping reduces hospitalization rates results from the MM-WES (Medco-Mayo Warfarin Effectiveness study). J Am Coll Cardiol. 2010 Jun 22;55(25):2804-12. doi: 10.1016/j.jacc.2010.03.009. Epub 2010 Apr 8. PMID 20381283
- [Background] Wang L, McLeod HL, Weinshilboum RM. Genomics and drug response. N Engl J Med. 2011 Mar 24;364(12):1144-53. doi: 10.1056/NEJMra1010600. No abstract available. PMID 21428770
- [Background] Aronson JK. Adverse drug reactions--no farewell to harms. Br J Clin Pharmacol. 2007 Feb;63(2):131-5. doi: 10.1111/j.1365-2125.2006.02860.x. No abstract available. PMID 17274787
- [Background] Edwards IR, Aronson JK. Adverse drug reactions: definitions, diagnosis, and management. Lancet. 2000 Oct 7;356(9237):1255-9. doi: 10.1016/S0140-6736(00)02799-9. PMID 11072960
- [Background] Gage BF, Eby C, Johnson JA, Deych E, Rieder MJ, Ridker PM, Milligan PE, Grice G, Lenzini P, Rettie AE, Aquilante CL, Grosso L, Marsh S, Langaee T, Farnett LE, Voora D, Veenstra DL, Glynn RJ, Barrett A, McLeod HL. Use of pharmacogenetic and clinical factors to predict the therapeutic dose of warfarin. Clin Pharmacol Ther. 2008 Sep;84(3):326-31. doi: 10.1038/clpt.2008.10. Epub 2008 Feb 27. PMID 18305455
- [Background] International Warfarin Pharmacogenetics Consortium; Klein TE, Altman RB, Eriksson N, Gage BF, Kimmel SE, Lee MT, Limdi NA, Page D, Roden DM, Wagner MJ, Caldwell MD, Johnson JA. Estimation of the warfarin dose with clinical and pharmacogenetic data. N Engl J Med. 2009 Feb 19;360(8):753-64. doi: 10.1056/NEJMoa0809329. PMID 19228618
- [Background] Garcia DA, Lopes RD, Hylek EM. New-onset atrial fibrillation and warfarin initiation: high risk periods and implications for new antithrombotic drugs. Thromb Haemost. 2010 Dec;104(6):1099-105. doi: 10.1160/TH10-07-0491. Epub 2010 Sep 30. PMID 20886196
- [Background] Meckley LM, Gudgeon JM, Anderson JL, Williams MS, Veenstra DL. A policy model to evaluate the benefits, risks and costs of warfarin pharmacogenomic testing. Pharmacoeconomics. 2010;28(1):61-74. doi: 10.2165/11318240-000000000-00000. PMID 20014877
- [Background] Relling MV, Klein TE. CPIC: Clinical Pharmacogenetics Implementation Consortium of the Pharmacogenomics Research Network. Clin Pharmacol Ther. 2011 Mar;89(3):464-7. doi: 10.1038/clpt.2010.279. Epub 2011 Jan 26. PMID 21270786
- [Background] Gandhi TK, Weingart SN, Borus J, Seger AC, Peterson J, Burdick E, Seger DL, Shu K, Federico F, Leape LL, Bates DW. Adverse drug events in ambulatory care. N Engl J Med. 2003 Apr 17;348(16):1556-64. doi: 10.1056/NEJMsa020703. PMID 12700376
- [Background] Huhtakangas J, Tetri S, Juvela S, Saloheimo P, Bode MK, Hillbom M. Effect of increased warfarin use on warfarin-related cerebral hemorrhage: a longitudinal population-based study. Stroke. 2011 Sep;42(9):2431-5. doi: 10.1161/STROKEAHA.111.615260. Epub 2011 Jul 28. PMID 21799168